CLINICAL TRIAL: NCT05293899
Title: The Pathogenesis of Depression - Possible Autoimmune Mechanisms
Status: Recruiting | Type: Observational
Sponsor: HaEmek Medical Center, Israel (Other)
Responsible Party: Principal Investigator, Einat Mader, M.D, HaEmek Medical Center, Israel
Other Study IDs: 143-19EMC
Record Dates: First submitted 2022-03-15; First posted 2022-03-24 (Actual); Last update posted 2022-03-24 (Actual); Status verified 2022-03

CONDITIONS: Depression; Autoimmune Diseases
MeSH Terms: conditions — Depression; Autoimmune Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — 1. Blood samples will be collected for genetic investigation. We will collect 10 ml of whole blood in EDTA tubes. The tubes will be refrigerated in 4-degree Celsius and will be delivered to the genetics laboratory in Ha Emek Medical Center. DNA will be then extracted from the samples and will be stored in the refrigerator. Genetics Laboratory, under the responsibility of Dr. Morad Khayat, the lab manager. After completion of the first phase proteome analysis, a further investigation into which genetic variants are most susceptible and those will be then analyzed. The information for each participant will be confidential for each patient and coded as noted.
  2. The genetic material will be kept for 10 years in the Genetic lab, for further investigation. Participants who will decide not to continue with the testing - their specimens will be destroyed.
  3. In any case of finding a known genetic aberration, the participants will be referred to genetic counseling.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: exome sequencing approach — Depending on the primary results in the proteomic and the metabolic profiling, this pilot study will search for genetic associations, using an exome sequencing approach to individuals. The findings will be compared to individuals without depression, and to relatives of depressed patients who suffer from autoimmune diseases.

SUMMARY:
It has long been claimed that depression, and other psychiatric illness, might be a manifestation of immune dysregulation involving the Central nervous system. Depression is associated with a significantly increased risk of autoimmune disease compared to those without a history of depression. The increased risk of autoimmune diseases is during the first year following the onset of depression .Conversely, up to 50% of patients with autoimmune diseases show an impairment of health-related quality of life and exhibit depressive symptoms.

The aggregation of depression and some specific autoimmune diseases may demonstrate shared inherited pathogenesis.

The first phase of the study will include patients with the diagnosis of depression. The control group will consist of a healthy population, according to medical records and will be recruited through a recruitment ad and volunteers. In the second phase of the study first and second-degree relatives (parents, siblings, children, grandparents, aunts, uncles and cousins) who are diagnosed with autoimmune disease/s will be recruited. Auto-immune diseases will include - Rheumatoid Arthritis (RA), juvenile idiopathic arthritis JIA), Seronegative spondyloarthropathies (SPA) including inflammatory bowel disease (IBD), psoriatic arthritis (PsA), and ankylosing spondylitis. Other autoimmune diseases: Systemic Lupus Erythematosus, Sjogren' syndrome (SS), systemic sclerosis (SSc), inflammatory myopathies (IIM), any Overlap of the above including mixed connective tissue disease (MCTD), systemic vasculitis (see Chapel Hill classification criteria). All autoimmune diseases will be confirmed by an expert rheumatologist or an internist. Celiac disease, Diabetes Mellitus type I, autoimmune thyroiditis, autoimmune hepatitis will be confirmed by a gastroenterologist, endocrinologist or an internist.

ELIGIBILITY:
Inclusion Criteria:

* Patients must meet DSM-5 (Diagnostic and Statistical Manual of Mental Disorders) criteria for a diagnosis of depression.
* Sufficient knowledge of the Hebrew language
* A stabled mental state. If hospitalized, patients are scheduled for discharge based on clinical assessment of psychiatric symptoms.

Exclusion Criteria:

* Mental co-morbidity.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The first phase of the study will include patients with the diagnosis of depression. The control group will consist of a healthy population, according to medical records and will be recruited through a recruitment ad and volunteers. In the second phase of the study first and second-degree relatives (parents, siblings, children, grandparents, aunts, uncles and cousins) who are diagnosed with autoimmune disease/s will be recruited.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2022-02-15 (Actual); Primary Completion 2026-02-15 (Estimated); Study Completion 2026-04-15 (Estimated)

PRIMARY OUTCOMES:
1. Find genetic association or genetic basis to depression associated with autoimmune diseases | 1 day
  1. Find genetic association or genetic basis to depression associated with autoimmune diseases

CONTACTS AND LOCATIONS:
Locations (1):
- Haemek medical center, Afula, Israel